CLINICAL TRIAL: NCT01025050
Title: Intrastromal Presbyopia Correction by Means of a Femtosecond Laser
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Priv.-Doz. Dr. med. Mike P. Holzer, University Ophthalmic Clinic, Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0905
Record Dates: First submitted 2009-11-25; First posted 2009-12-03 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Presbyopia
Keywords: Presbyopia; Intrastromal; Femtosecond Laser; minimal-invasive; INTRACOR; Enhance Near Visual Acuity
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): In this group the smallest ring diameter will be applied.
  Interventions: Procedure: Intrastromal Correction of Presbyopia
- Group B (Experimental): In this group the intermediate ring diameter will be applied.
  Interventions: Procedure: Intrastromal Correction of Presbyopia
- Group C (Experimental): In this group the biggest ring diameter will be applied.
  Interventions: Procedure: Intrastromal Correction of Presbyopia

INTERVENTIONS:
Procedure: Intrastromal Correction of Presbyopia — On all patients an intrastromal pattern consisting of concentric rings will be applied.

SUMMARY:
This clinical study is an open, prospective, multi-centre eye study consisting of three study arms to determine the safety and efficacy of intrastromal incisions for the correction of visual acuity on presbyopic eyes. The hypothesis of the study is that by means of intrastromal incisions, near visual acuity can be improved in presbyopic eyes in a safe and effective way.

DETAILED DESCRIPTION:
This clinical study is an open, prospective, multi-centre eye study consisting of three study arms to determine the safety and efficacy of intrastromal incisions for the correction of visual acuity on presbyopic eyes. The incisions are applied by means of the FEMTEC femtosecond laser system with the INTRACOR software module using patterns consisting of 6 concentric rings and 3 different inner ring diameters. A similar pattern with 5 concentric rings and only one fixed inner diameter is currently under clinical investigation.

The hypothesis of the study is that by means of intrastromal incisions, near visual acuity can be improved in presbyopic eyes in a safe and effective way.

The intrastromal incisions are performed by the femtosecond laser FEMTEC, which is CE certified for various therapeutic indications. The incision eliminates both an epithelial and an endothelial opening of the cornea whereby the minimally invasive character of this form of treatment is guaranteed. A detailed pre-operative examination will ensure that every interested and willing patient fulfils the inclusion criteria of this study. Post-operative examinations, which should document the success of the treatment, are to be carried out after 24 hours, 1 week, 1 month, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18 years old
* Patients must have read, understood and signed the Patient Information
* Patients are willing and able to return for follow-up examinations
* Stable distance refraction
* Manifested Refraction (see Table 1 for more details) :

  * Cylinder: -0.5 D to 0 D
  * Sphere: 0.25 D to 1.25 D
  * Spherical equivalent: Minimum 0.25 D
* Best corrected distance visual acuity of the eye to be treated at least 0.8
* Subjects must have presbyopia as determined by an age-related need for optical aid (≥ +1.5 D) for reading with their best distance correction.

Exclusion Criteria:

* Minimum cornea thickness < 500 µm
* Ocular dominance (only non-dominant eyes should be included)
* Uncorrected Near Visual Acuity of 0.5 or better
* Difference between manifested and cycloplegic refraction of > 0.75 D in spherical equivalent
* Median K values < 40 D or > 46 D
* Topographical astigmatism > 5 D
* Abnormal corneal topography
* Patients with previous corneal operations on the eye to be treated (e.g. LASIK, PRK, X-Linking; this does not include cataract operations)
* Scarring or opacity of the cornea
* Transplanted cornea
* Connective tissue weaknesses
* Keratectasia and other diseases of the cornea
* Patients with wound-healing disorders such as connective tissue disease, autoimmune illnesses, immunodeficiency illnesses, ocular herpes zoster or simplex, endocrine diseases, lupus, rheumatoid arthritis
* Patients regularly taking medicines that could influence the result of the treatment
* Glaucoma or a risk of glaucoma
* Patients with concentration disorders, epilepsy, diabetes mellitus and other complicating diseases
* Patients with disorders of the ocular muscle, such as nystagmus or strabismus
* Sensitivities to the drugs used in this study
* Continual wearing of contact lenses before the pre-examination and before the operation. Patients must refrain from wearing contact lenses for at least 14 days prior to these dates
* Patients who are pregnant or are lactating
* Patients who are participating in another ophthalmological clinical study
* Best corrected distance visual acuity of the second, not to be treated eye is 0.5 or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-12; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The proportion of treated eyes who gained uncorrected near visual acuity of at least 2 lines. This proportion should be greater than 70%. | 6 months follow up

SECONDARY OUTCOMES:
The proportion of treated eyes that lose more than two lines of best corrected visual acuity (BSCVA). This proportion should be no greater than 5 %. | 6 months follow up

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - University Eye Clinic Heidelberg, Heidelberg, Baden-Wurttemberg
  - FreeVis LASIK Center Mannheim GmbH, Mannheim, Baden-Wurttemberg
  - Augenklinik am Marienplatz AG & Co. KG, Munich, Bavaria
  - Eye-clinic for Refractive and Ophthalmo-Surgery, EJK Niederrhein, Duisburg, North Rhine-Westphalia

REFERENCES:
- [Derived] Thomas BC, Fitting A, Khoramnia R, Rabsilber TM, Auffarth GU, Holzer MP. Long-term outcomes of intrastromal femtosecond laser presbyopia correction: 3-year results. Br J Ophthalmol. 2016 Nov;100(11):1536-1541. doi: 10.1136/bjophthalmol-2015-307672. Epub 2016 Feb 22. PMID 26903524